CLINICAL TRIAL: NCT03863912
Title: Impact of Disney Movies During Chemotherapy on QOL of Gynecologic Oncology Patients: A Prospective Study
Brief Title: Impact of Disney Movies During Chemotherapy on QOL of Gynecologic Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Sophie Pils, MD, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1908/2017
Record Dates: First submitted 2019-02-25; First posted 2019-03-05 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Ovarian Cancer; Chemotherapy; Quality of Life
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disney (Active Comparator): watch Disney movies and fill out EORTC QLQ-C30 (Version 3) and EORTC QLQ-FA12 surveys
  Interventions: Other: Disney movie; Other: EORTC QLQ-C30 and EORTC QLQ-FA12 surveys
- Control (Other): fill out EORTC QLQ-C30 (Version 3) and EORTC QLQ-FA12 surveys
  Interventions: Other: EORTC QLQ-C30 and EORTC QLQ-FA12 surveys

INTERVENTIONS:
Other: Disney movie — Disney movie on portable DVD Player.
  Arms: Disney
Other: EORTC QLQ-C30 and EORTC QLQ-FA12 surveys — EORTC QLQ-C30 and EORTC QLQ-FA12 surveys

SUMMARY:
To evaluate the impact of Disney movies on quality of life (QOL) of gynecologic oncology patients.

25 Patients are watching Disney movies on portable DVD players during chemotherapy, 25 patients are not allowed to watch TV.

EORTC QLQ-C30 and EORTC QLQ-FA12 surveys are given to the patients before and after the six chemotherapies.

Hypothesis: Disney movies can elevate patients QOL.

ELIGIBILITY:
Inclusion Criteria:

* planned 6 cycles of chemotherapy with carboplatin/paclitaxel or carboplatin/pegylated liposomal doxorubicin
* Age >18 years

Exclusion Criteria:

* inadequate knowledge of the German language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only gynecological cancer patients are included
Enrollment: 56 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2018-11-29 (Actual)

PRIMARY OUTCOMES:
Change of Quality of life during 6 cycles of chemotherapy | Measured before and after each chemotherapy (at baseline and on average after 3, 6, 9, 12, 15 weeks after inclusion in patients with carboplatin/paclitaxel or after 4, 8, 12, 16, 20 weeks after inclusion in patients with carboplatin/doxorubicin)
  To compare change in Quality of Life, as defined by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30 (Version 3)) during 6 cycles of chemotherapy.
  The EORTC QLQ-C30 (Version 3) uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.
  The EORTC QLQ-C30 (Version 3) uses for the questions 29 and 30 a 7-points scale. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. First of all, raw score has to be calculated with mean values. Afterwards linear transformation is performed to be comparable. More points are considered to have a better outcome.
Change of Fatigue during 6 cycles of chemotherapy | Measured before and after each chemotherapy (at baseline and on average after 3, 6, 9, 12, 15 weeks after inclusion in patients with carboplatin/paclitaxel or after 4, 8, 12, 16, 20 weeks after inclusion in patients with carboplatin/doxorubicin)
  To compare change in Fatigue, as defined by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Fatigue (EORTC QLQ-FA12) during 6 cycles of chemotherapy.
  The EORTC QLQ-FA12 uses for the questions 1 to 12 a four-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome. Raw score has to be calculated using the mean value for the questions 1 to 12.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Pils, MD, Principal Investigator — Medical University of Vienna, Department of General Gynecology and Gynecologic Oncology
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pils S, Ott J, Reinthaller A, Steiner E, Springer S, Ristl R. Effect of Viewing Disney Movies During Chemotherapy on Self-Reported Quality of Life Among Patients With Gynecologic Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2020 May 1;3(5):e204568. doi: 10.1001/jamanetworkopen.2020.4568. PMID 32391894